CLINICAL TRIAL: NCT03730844
Title: Functional Outcomes in Children Post Critical Illness
Status: Completed | Type: Observational
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2014/2073
Record Dates: First submitted 2018-10-25; First posted 2018-11-05 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2018-10

CONDITIONS: Critical Illness
Keywords: Functional outcomes; Skeletal muscle
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Critically ill children: Children admitted to the PICU.
- Healthy controls: Healthy controls, not admitted to the PICU, without pre-existing medical conditions.

SUMMARY:
Improvements in medical care have led to decreasing mortality rates in critically ill children, which have been reported to be as low as 5%. However, surviving critical illness does not necessarily translate to a return to pre-critical illness functional and developmental levels. Adult literature has shown that critical illness increases functional disability for up to five years post intensive care unit stay. We hypothesize that children experience similar functional disabilities as a result of critical illness, which may, as in adults, be primarily due to muscle wasting. The aim of this prospective observational pilot study is establish the relationship between intensive care unit stay and functional outcomes in pediatric survivors of critical illness.

DETAILED DESCRIPTION:
Background:

Mortality rates in critically ill children have decreased significantly in recent years, with current rates reported to be as low as 5%. However, increased survival may result in significant morbidity. Herridge et al. demonstrated that adults admitted to the intensive care unit (ICU) for acute respiratory distress syndrome experienced functional disability which persisted up to 5 years after their ICU stay. There now exists a substantial body of literature that adult critical care survivors suffer significant impairment in their quality of life, which is a growing public health issue.

In critically ill children, Namachivayam et al. showed that among children with pediatric intensive care unit (PICU) stay > 28days, 34% of survivors had an unfavourable functional outcome (defined as moderate or severe disability with dependence on others for care as measured by the Glasgow Outcome Scale). Health related quality of life was also affected, with 68% of survivors having poorer quality of life scores as measured by the Health State Utilities Index. Thus, clinicians have argued that mortality may not be the most meaningful outcome measure for PICU patients. Alternative outcome measures such as functional status and quality of life of children post critical illness may give a better overall assessment of how well children cope with surviving critical illness, and how their normal development is affected.

In adults there is a growing understanding of the burden of critical care survivors on families and caregivers. Limited data exists regarding the families and caregivers of survivors of pediatric critical illness, and local data is lacking.

Aim:

The investigator's aim is to assess the impact of critical illness on functional outcomes in survivors of pediatric critical illness, as well as the impact on the caregivers.

Hypotheses:

1. Children surviving critical illness demonstrate significant functional impairment that persists for up to 12 months.
2. Caregivers of children surviving critical illness experience prolonged lower quality of life and significant economic stress.
3. Low muscle mass secondary to muscle wasting is highly associated with said functional disability.

Specific objectives:

1. To describe short and long term functional outcomes in pediatric survivors.
2. To describe the relationship between muscle wasting and functional outcome measures.
3. To elucidate the relationship between pediatric critical illness survivor functional outcomes and caregiver's long term quality of life and lost workdays.
4. To establish the relationship between in-PICU and in-hospital nutrition and physical activity and functional outcomes after a year.

ELIGIBILITY:
Critically ill children group

Inclusion Criteria:

* Anticipated at least 48 hours of PICU stay
* At least 1 organ dysfunction
* Expected to survive to PICU discharge

Exclusion Criteria:

* Amputations
* Pre-existing progressive neuromuscular disease
* Oncological disease
* Premature infants, before corrected gestational age 1 month

Healthy controls group

Inclusion criteria:

* No pre-existing medical condition requiring active treatment

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Critically ill children will be recruited during their PICU stay at KK Women's and Children's Hospital. They will be followed throughout their PICU stay, at hospital discharge, and 6-12 months post discharge.
  Healthy controls will be recruited from the general public by word of mouth. They will undergo assessments at a single time-point.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2015-04-13 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change in functional status | PICU discharge (expected average 7 days from admission), hospital discharge (expected average 17 days from PICU admission), 6-12 months post discharge
  Change in Functional Status Scale (FSS) scores from baseline

SECONDARY OUTCOMES:
Change in functional status | Hospital discharge (expected average 17 days from PICU admission), 6-12 months post discharge
  Change in functional status from baseline, as measured by the Pediatric Evaluation of Disability Inventory - computer adaptive test (PEDI-CAT).
Rectus femoris cross-sectional area | Baseline, Day 3, 7, 10 of PICU stay, PICU discharge (expected average 7 days from admission), hospital discharge (expected average 17 days from PICU admission), 6-12 months post discharge
  Change in cross-sectional area of the rectus femoris measured by ultrasonography from baseline and in comparison to healthy controls
Health related quality of life: Pediatric Quality of Life Inventory (PedsQL) 4.0 generic module and Infant scales | PICU discharge (expected average 7 days from admission), hospital discharge (expected average 17 days from PICU admission), 6-12 months post discharge
  Patient or proxy-reported health related quality of life measured using the age appropriate PedsQL 4.0 generic module (2 - 18 years) and the PedsQL Infant scales (0 - 24 months). Total scores will be calculated on a scale of 0 - 100 (with 100 being the best possible score).
Caregiver health related quality of life | Hospital discharge (expected average 17 days from PICU admission), 6-12 months post discharge
  Parental health-related quality of life measured using the 36-Item Short Form Health Survey (SF-36) questionnaires. SF-36 mental component summary scores (MCS) and physical component summary scores (PCS) will be reported on a scale of 0 - 100 (with 100 being the best possible score).
Hand grip strength | Hospital discharge (expected average 17 days from PICU admission), 6-12 months post discharge
  Hand grip strength test in children 6 years and above, compared to healthy controls

OTHER OUTCOMES:
24-hour dietary recall | 6-12 months post discharge
  Nutritional intake assessed by 24-hour dietary recall

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ong C, Lee JH, Wong JJM, Leow MKS, Puthucheary ZA. Skeletal Muscle Changes, Function, and Health-Related Quality of Life in Survivors of Pediatric Critical Illness. Crit Care Med. 2021 Sep 1;49(9):1547-1557. doi: 10.1097/CCM.0000000000004970. PMID 33861558